CLINICAL TRIAL: NCT00531648
Title: The System of Relationships Between Parents and Their Toddlers, With Eating Disorders and Sensory Processing Disorders Within Meal and Play Situations
Brief Title: Relationships Between Toddlers With Feeding Disorder and SPD and Their Parents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Other Study IDs: Feeding disorder-33CTIL
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2007-09

CONDITIONS: Feeding and Eating Disorders of Childhood; Developmental Disabilities
Keywords: Toddlers that having feeding disorders and SPD
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Families with toddlers that having feeding disorders and SPD

SUMMARY:
The researched attends to observe the relationships between toddlers that were diagnosed as SPD and as having feeding disorder (by DSM-R-IV)and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Toddlers aged between one year to two and a half years
* Toddlers diagnosed as SPD by occupational therapist
* Toddlers diagnosed as having feeding disorder by psychiatric physician according to DSM-R-IV
* Toddlers that are normally developed as reported by pediatrician

Exclusion Criteria:

* Compliant families
* Toddlers with poor health

Ages: 12 Months to 30 Months | Sex: All
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2007-09; Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Irit Orian, M.D., Principal Investigator — Mental health unit for preschoolers, Ashdod, Israel; Inbal Heimann, B.A., Study Director — Mental health unit for preschoolers, Ashdod, Israel
Locations (1):
- Mental health unit for preschoolers, Ashdod, Israel